CLINICAL TRIAL: NCT06740695
Title: The Effect of Health Belief Model-Based Education Given to Pregnant Women Via WhatsApp on Self-Efficacy and Risk Perception in Pregnancy in Gestational Diabetes
Brief Title: Health Belief Model Based Education for Pregnant Women With Gestational Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Mine Gokduman Keles, Burdur Mehmet Akif Ersoy University DOCTORATE LECTURER MIDWIFERİY, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/12 GO 2024/800
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Complications
Keywords: Health Belief Model Gestational Diabetes Self-efficacy risk perception
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Education group (Active Comparator)
  Interventions: Behavioral: Education group

INTERVENTIONS:
Behavioral: Education group — The training materials were prepared in line with the researchers and expert opinions were obtained. Trainings will be given for two weeks. After the trainings are completed, reminder information will be sent to the pregnant women via text messages every other day to inform them that the trainings are continuing. Reminder information prepared as text messages will be sent to the pregnant women's mobile phones. 4 weeks after the first training, the same training will be reminded again via WhatsApp as a summary training by emphasizing key points.
  The trainings will be carried out by an expert researcher in the field. In the training content prepared in line with WhatsApp, the risks that may be seen during pregnancy and Gestational Diabetes Mellitus;
  * Sensitivity perception and Seriousness perception, perceived risks that may be seen during pregnancy
  * Health motivation perception, the pregnant woman's beliefs and practices regarding being healthy,
  * Benefit perception, pregnancy follow
  Arms: Education group

SUMMARY:
Gestational diabetes (GDM) is a type of diabetes that occurs as a result of intolerance of carbohydrate metabolism during pregnancy in an individual whose blood glucose concentration is within normal limits before pregnancy. GDM is an important condition that should be handled carefully. Because it is one of the most common metabolic diseases during pregnancy and poses risks to the health of the mother, fetus and newborn. Increasing Self-Efficacy in Gestational Diabetes with education based on the Health Belief Model,

DETAILED DESCRIPTION:
Gestational diabetes (GDM) is a type of diabetes that occurs as a result of intolerance of carbohydrate metabolism during pregnancy in an individual whose blood glucose concentration is within normal limits before pregnancy. GDM is an important condition that should be addressed carefully. Because it is one of the most common metabolic diseases during pregnancy and brings risks to the health of the mother, fetus and newborn. The prevalence of GDM is 1-14% without considering geographical changes, and the incidence of Type 2 diabetes diagnosed at the end of pregnancy increases with the increase in the rate of occurrence in fertile obese women. Similar to Type 2 diabetes, the main problem in gestational diabetes is that production is not sufficient for the need due to insulin resistance. In addition to the fact that consuming more calories than normal due to uncontrolled nutrition, increasing the fat rate in the body and exercise and lack of movement are important factors in the emergence of gestational diabetes, hormones such as cortisol, prolactin, human placental lactogen, progesterone, which have an adverse effect on insulin, and placental insulinase enzymes that accelerate insulin destruction also play a major role in the emergence of gestational diabetes. Regardless of the main problem or the type of diabetes, pregnancy complications are related to the degree to which blood glucose cannot be controlled. Pregnancy-related diabetes complications generally consist of two groups. The first group consists of congenital anomalies that occur due to metabolic conditions in the first trimester of pregnancy. A significant increase in blood glucose in the first trimester of pregnancy is one of the most important teratogenic factors. It is reported that approximately 27% of pregnant women with uncontrolled high glucose in the first trimester develop congenital anomalies. It is stated in the literature that providing effective education to individuals with gastrointestinal diabetes facilitates the control of complications that may occur due to diabetes. In addition, the absence of such a study in the literature suggests that our study will make a very good contribution to the literature.To increase self-efficacy in gestational diabetes through training based on the Health Belief Model,

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,

  * In the second trimester,
  * Primiparous,
  * Have adequate communication skills,
  * Literate,
  * Can read and understand Turkish,
  * Recently diagnosed with GDM,
  * Have a singleton pregnancy,
  * Pregnant women who agree to participate in the study will be included.
  * Continuing pregnancy school

Exclusion Criteria:

* Pregnant women with risky pregnancies,

  * Multiple pregnancies were not included in the study.
  * Pregnant women with previous type 1 or type 2 diabetes,
  * Have a psychiatric diagnosis,
  * Have a physical disability,
  * Have communication problems will be excluded.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Risk Perception Scale (GRP) | 1 HOUR
  The scale was developed by Heaman and Gupton (2009) to assess the risk perception of pregnant women. The Turkish validity and reliability study of the scale was conducted by Evcili and Dağlar (2019) . The risk perception scale consists of 9 items and 2 sub-dimensions. The scale is a visual analog measurement tool. The scale consists of 9 items and 2 factors. There is a 0-100 mm linear line immediately below each item in the scale, indicating "no risk" and "extremely high risk". The total score of the scale is found by adding the scores for each of the nine items and dividing the obtained score by 9. A score can also be made for the factors of the scale: The score for the "Risk perception of the pregnant woman towards her baby" factor is found by adding the scores for each of the 5 items under this factor and dividing the obtained score by 5. The score for the "Risk perception of the pregnant woman towards herself" factor is obtained by add
Self-Efficacy Scale in Gestational Diabetes (GESGD): | 1 HOUR
  Developed by Polat and Avdal (2020), the Self-Efficacy Scale in Gestational Diabetes is a five-point Likert-type scale consisting of 23 items and four sub-dimensions. The total Cronbach alpha value of the scale was determined as 0.654. Its sub-dimensions are Diet and Weight Management, Complication Precautions, Nutrition Education Compliance and Medical Treatment Applications. It has been emphasized that as the score to be obtained from the scale increases as a result of the coding of the positive and negative expressions in the scale, the individual's self-efficacy will increase and that he/she will be able to effectively perform his/her own care as a result of the training he/she receives.

IPD SHARING:
Plan to Share IPD: No